CLINICAL TRIAL: NCT07200557
Title: Reassessing the Role of Routine Radiographs After Spinal Fusion Surgery
Acronym: RRASP
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S68783
Record Dates: First submitted 2025-09-10; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Radiography; Spinal Fusion
Keywords: Routine radiographs; Spinal fusion; Clinical utility; Spinal fusion surgery; Radiographs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing spinal fusion surgery (2011-2021) at University Hospitals Leuven: Retrospective cohort of adult patients (≥18 years) who underwent spinal fusion surgery for degenerative spinal conditions at University Hospitals Leuven between 2011 and 2021. Patients were followed for at least 12 months after surgery, with data collected from postoperative follow-up visits, including clinical course, radiographic findings, and subsequent management decisions.

SUMMARY:
Routine radiographs are commonly obtained after spinal fusion surgery to monitor postoperative evolution and detect complications. However, the actual contribution of these radiographs to clinical decision-making remains unclear. This retrospective cohort study evaluates the frequency and clinical impact of routine postoperative radiographs in patients undergoing spinal fusion surgery at University Hospitals Leuven.

DETAILED DESCRIPTION:
Routine radiographs are commonly obtained after spinal fusion surgery to assess implant position, fusion progress, and potential complications. Yet, their actual contribution to patient care remains uncertain, and routine use may expose patients to unnecessary radiation and increase healthcare costs.

In this retrospective cohort study, the investigators will evaluate the clinical utility of routine radiographs during the first postoperative year after spinal fusion surgery at University Hospitals Leuven (2011-2021).

The investigators will review each follow-up visit to record the clinical course, radiographic findings, and whether these influenced further diagnostic tests or therapeutic interventions.

The investigators will primarily assess how often radiographs lead to a change in management. Secondary analyses will determine the proportion of abnormal versus normal radiographs, the relationship between clinical course and imaging results, and whether demographic or surgical factors predict radiographic utility.

By analyzing nearly 1,000 patients and more than 2,800 visits, the investigators will provide one of the most comprehensive evaluations of routine postoperative radiographs to date, aiming to guide more efficient, evidence-based follow-up strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent spinal fusion surgery at UZ Leuven, including the cervical, thoracic and lumbar spine for a degenerative condition
* Adults of 18 years and older
* Follow up at least 3 months after surgery

Exclusion Criteria:

* Non-degenerative (kypho) scoliosis
* Indications other than degenerative conditions and (adult) isthmic spondylolisthesis (e.g. tumor, septic arthritis, trauma,…)
* Chronic neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spinal fusion surgery (2011-2021) for degenerative conditions at University Hospitals Leuven
Sampling Method: Non-Probability Sample
Enrollment: 978 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of radiographs that led to further diagnostic tests or therapeutic interventions within 12 months post-surgery | Within 12 months after spinal fusion surgery
  Percentage of follow-up visits with routine radiographs in which the radiograph resulted in further diagnostic testing (e.g., CT, MRI) or a therapeutic intervention (e.g., medication change, reoperation).

SECONDARY OUTCOMES:
Proportion of abnormal versus normal radiographs | Within 12 months after spinal fusion surgery
  Percentage of routine postoperative radiographs classified as abnormal compared to those classified as normal, based on radiologist or surgeon interpretation.
Correlation between clinical course and management decisions | Within 12 months after spinal fusion surgery
  Percentage of follow-up visits in which the patient was symptomatic versus asymptomatic, compared to the percentage of those visits that resulted in further diagnostic testing or therapeutic intervention.
Correlation of demographic factors with radiographic utility | Within 12 months after spinal fusion surgery
  Percentage of radiographs leading to additional diagnostic tests or therapeutic interventions, stratified by demographic variables (age in years, sex, body mass index in kg/m²).
Correlation of surgical factors with radiographic utility | Within 12 months after spinal fusion surgery
  Percentage of radiographs leading to additional diagnostic tests or therapeutic interventions, stratified by surgical variables (fusion level: cervical, thoracic, lumbar; number of fused segments; type of instrumentation).

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Rummens, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
This is a retrospective, single-center study. No individual participant data will be made publicly available. Summary results will be reported in peer-reviewed publications.